CLINICAL TRIAL: NCT02224469
Title: Utrecht Neural Prosthesis (UNP): A Pilot Study on Controllability of Brain Signals and Application in locked-in Patients
Brief Title: First Study With a Brain Implant to Help Locked-in Patients Communicate at Home
Acronym: UNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Erik Aarnoutse, PhD, Study Coordinator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCU 12-370; STW 12803 (Other Grant/Funding Number: Technology Foundation STW)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Locked-In Syndrome
Keywords: Brain-Computer Interface; Motor Cortex; Dorsolateral Prefrontal Cortex; Quality of Life
MeSH Terms: conditions — Locked-In Syndrome | interventions — Electrocorticography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECoG (electrocorticography) sensing (Experimental): Use ECoG-based Brain Computer interface to control assistive technology
  Interventions: Device: ECoG (electrocorticography) sensing

INTERVENTIONS:
Device: ECoG (electrocorticography) sensing — Implant electrodes and sensing device and use for control of Assistive Technology
  Other Names: Activa PC + S

SUMMARY:
In this study a new means of communication for people with locked-in syndrome will be tested. The investigators will record brain signals directly from the surface of the brain by means of a completely implantable system. These brain signals are fed wirelessly into an assistive technology device and will control this device for communication and environmental control at the users home.

DETAILED DESCRIPTION:
In this pilot study we will provide locked-in people with a new means of communication which has not been possible up to now. For the first time, we will test whether we can record and decode neural signals obtained directly from the brain, for control over a computer. The target population is people with locked-in syndrome. For these patients there is no technique available to allow them to communicate unaided. We have developed a brain-computer interface (BCI) system that can read activity directly from the brain, and can convert the activity to a digital switch. The system, called the Utrecht Neural Prosthesis (UNP), consists of an implantable amplifier for electrical brain signals, a set of electrodes positioned on the surface of the brain and a wireless receiver, placed outside of the body. A dedicated computer will convert the signals to electrical pulses for standard Assistive Technology devices. The UNP can in principle enable the patient to engage in any activity that is offered by commercial Assistive Technology companies that can be performed with switch signals, for instance operating home apparatus or writing text. Most importantly, we aim to achieve unsupervised function of the BCI, meaning that the patient will be able to use it at home without the aid of researchers or other experts (but with minimal caregiver assistance).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75
* Locked-in status (i.e. severely paralyzed with communication problems)

  * in case of trauma or stroke: at least 1 year after the event
  * in case of a neuromuscular disease: slow progression allowed
* Rudimentary form of communication possible (e.g. through assistive technology, eye blinks or eye movements, severely impaired speech)
* Mentally and physically capable of giving informed consent
* Lives in or close to the Netherlands
* MR compatible

  * able to lie flat in the scanner
  * no metal objects in or attached to the body
  * no claustrophobia
* Visus (largely) intact
* Cognition intact (IQ>80)
* Compatible with implantation procedure

  * good respiratory function or stable respiratory situation using ventilation assistance

Exclusion Criteria:

* Strong and frequent spasms
* Vital indication for blood thinners
* Current brain tumor or history of tumor resection
* Quick medical or neurological deterioration
* Patients who are considered legally incapable (and who therefore will not be able to give informed consent)
* Current or recent psychiatric disorder
* Catabolic state
* Allergy to the materials of the implant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick F Ramsey, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
selected datasets will be available through a public repository after publication of results
Time Frame: From Nov 14, 2016, no end date
Access Criteria: According to http://datadryad.org/pages/policies
URL: http://datadryad.org/resource/doi:10.5061/dryad.k9f10

REFERENCES:
- [Background] Vansteensel MJ, Hermes D, Aarnoutse EJ, Bleichner MG, Schalk G, van Rijen PC, Leijten FS, Ramsey NF. Brain-computer interfacing based on cognitive control. Ann Neurol. 2010 Jun;67(6):809-16. doi: 10.1002/ana.21985. PMID 20517943
- [Background] Torres Valderrama A, Paclik P, Vansteensel MJ, Aarnoutse EJ, Ramsey NF. Error probability of intracranial brain computer interfaces under non-task elicited brain states. Clin Neurophysiol. 2012 Dec;123(12):2392-401. doi: 10.1016/j.clinph.2012.05.006. Epub 2012 Jun 12. PMID 22695047
- [Result] Vansteensel MJ, Pels EGM, Bleichner MG, Branco MP, Denison T, Freudenburg ZV, Gosselaar P, Leinders S, Ottens TH, Van Den Boom MA, Van Rijen PC, Aarnoutse EJ, Ramsey NF. Fully Implanted Brain-Computer Interface in a Locked-In Patient with ALS. N Engl J Med. 2016 Nov 24;375(21):2060-2066. doi: 10.1056/NEJMoa1608085. Epub 2016 Nov 12. PMID 27959736
- [Result] Freudenburg ZV, Branco MP, Leinders S, van der Vijgh BH, Pels EGM, Denison T, van den Berg LH, Miller KJ, Aarnoutse EJ, Ramsey NF, Vansteensel MJ. Sensorimotor ECoG Signal Features for BCI Control: A Comparison Between People With Locked-In Syndrome and Able-Bodied Controls. Front Neurosci. 2019 Oct 16;13:1058. doi: 10.3389/fnins.2019.01058. eCollection 2019. PMID 31680806
- [Result] Pels EGM, Aarnoutse EJ, Leinders S, Freudenburg ZV, Branco MP, van der Vijgh BH, Snijders TJ, Denison T, Vansteensel MJ, Ramsey NF. Stability of a chronic implanted brain-computer interface in late-stage amyotrophic lateral sclerosis. Clin Neurophysiol. 2019 Oct;130(10):1798-1803. doi: 10.1016/j.clinph.2019.07.020. Epub 2019 Jul 27. PMID 31401488
- [Result] Pels EGM, Aarnoutse EJ, Ramsey NF, Vansteensel MJ. Estimated Prevalence of the Target Population for Brain-Computer Interface Neurotechnology in the Netherlands. Neurorehabil Neural Repair. 2017 Jul;31(7):677-685. doi: 10.1177/1545968317714577. Epub 2017 Jun 22. PMID 28639486
- [Result] Leinders S, Vansteensel MJ, Branco MP, Freudenburg ZV, Pels EGM, Van der Vijgh B, Van Zandvoort MJE, Ramsey NF, Aarnoutse EJ. Dorsolateral prefrontal cortex-based control with an implanted brain-computer interface. Sci Rep. 2020 Sep 22;10(1):15448. doi: 10.1038/s41598-020-71774-5. PMID 32963279
- [Result] Leinders S, Vansteensel MJ, Piantoni G, Branco MP, Freudenburg ZV, Gebbink TA, Pels EGM, Raemaekers MAH, Schippers A, Aarnoutse EJ, Ramsey NF. Using fMRI to localize target regions for implanted brain-computer interfaces in locked-in syndrome. Clin Neurophysiol. 2023 Nov;155:1-15. doi: 10.1016/j.clinph.2023.08.003. Epub 2023 Aug 18. PMID 37657190
- [Result] Vansteensel MJ, Leinders S, Branco MP, Crone NE, Denison T, Freudenburg ZV, Geukes SH, Gosselaar PH, Raemaekers M, Schippers A, Verberne M, Aarnoutse EJ, Ramsey NF. Longevity of a Brain-Computer Interface for Amyotrophic Lateral Sclerosis. N Engl J Med. 2024 Aug 15;391(7):619-626. doi: 10.1056/NEJMoa2314598. PMID 39141854
- [Derived] Leinders S, Aarnoutse EJ, Branco MP, Freudenburg ZV, Geukes SH, Schippers A, Verberne MSW, van den Boom M, van der Vijgh B, Crone NE, Denison T, Ramsey NF, Vansteensel MJ. DO NOT LOSE SLEEP OVER IT: IMPLANTED BRAIN-COMPUTER INTERFACE FUNCTIONALITY DURING NIGHTTIME IN LATE-STAGE AMYOTROPHIC LATERAL SCLEROSIS. medRxiv [Preprint]. 2024 Oct 15:2024.10.11.24315027. doi: 10.1101/2024.10.11.24315027. PMID 39484239
- See also: Related Info for laymen — http://www.neuroprothese.nl
- See also: Info on research group — http://www.nick-ramsey.eu
- Available data/document: Individual Participant Data Set: k9f10 — http://datadryad.org/resource/doi:10.5061/dryad.k9f10

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ECoG (electrocorticography) sensing
Started | 6
Completed | 3
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | ECoG (Electrocorticography) Sensing
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reaching Proficiency Level 2: Unsupervised BCI Performance
Description: The system correctly detects a switch brain signal within 10 sec in a real life, cognitively engaging context, such as operating a spelling device. A formal test has been designed, in which the patient has to copy a 30 character sentence within 30 minutes, with a margin of 20% faulty characters.
Time Frame: up to 1 year
Population: This is analyzed in the participants who received an implant
Measure: Count of Participants; unit: Participants
Arm/Group | ECoG (electrocorticography) sensing
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Patient Device Satisfaction
Description: The Québec User Evaluation of Satisfaction with Assistive Technology (QUEST) 2.0, a self-report or interview-based scale, designed to evaluate a person's satisfaction with a wide range of assistive technology, consisting of a 12 questions scale from 1(very dissatisfied) - 4(very satisfied). Reported is mean score. Higher scores are better.
Time Frame: 8 years
Population: participant with home use
Measure: Number; unit: score on a scale
Arm/Group | ECoG (electrocorticography) sensing
Number analyzed (Participants) | 1
score on a scale | 3.5

3. Secondary Outcome: Effects Device on Quality of Life
Description: Psychosocial Impact of Assistive Devices Scale (PIADS), a 26-item, self-report questionnaire designed to assess the effects of an assistive device on functional independence, well-being, and quality of life. Score range is -3 to 3, larger values indicate a more positive effect of the device. Outcome is averaged over three domains (competence, adaptability, and self-esteem)
Time Frame: 3 years
Population: participant with home use
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | ECoG (electrocorticography) sensing
Number analyzed (Participants) | 1
score on a scale | 2.43 [-2 to 3]

4. Secondary Outcome: Quality of Life by Scoring Subjective Well-being in ACSA Score
Description: Anamnestic Comparative Self-Assessment (ACSA), a self-anchoring rating scale for subjective well-being score, ranges from -5 (worst period in life) to +5 (best period in life). Higher scores are a better outcome.
Time Frame: 4.5 years
Population: participant with home use
Measure: Number; unit: score on a scale
Arm/Group | ECoG (electrocorticography) sensing
Number analyzed (Participants) | 1
score on a scale | 2

5. Secondary Outcome: Hours of Use of BCI Device Per Day
Description: The hours of use of the BCI device as determined by logging within the home use software. Only hours of use with full featured home use software and appropriate signal amplitude. The period where signal amplitude declined, possibly due to participants disease progression, is not taken into account.
Time Frame: Time frame starts when participant receives a system with the full feature set for 24h home use and ends when signal decline starts influencing hours of use per day, an average of 1 year
Population: participant with home use
Measure: Mean (Full Range); unit: hours per day
Arm/Group | ECoG (electrocorticography) sensing
Number analyzed (Participants) | 1
hours per day | 21.26 [19 to 23.5]

6. Other Pre Specified Outcome: Supervised BCI Performance
Description: The patient is able to generate switch commands with at least 80 % correct, with the help of a BCI researcher and/or caregiver (using a formal test)
Time Frame: up to 28 weeks
Population: only participants that received an implant
Measure: Count of Participants; unit: Participants
Arm/Group | ECoG (electrocorticography) sensing
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 8.5 years
Arm/Group | ECoG (electrocorticography) sensing
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECoG (electrocorticography) sensing (N=6)
fever (Infections and infestations) | 1 (1) — 1 day readmission in hospital after surgery
disease related respiratory failure (Nervous system disorders) | 2 (2) — death before implantation
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — hospitalisation due to pneumonia
low oxygen (Respiratory, thoracic and mediastinal disorders) | 1 (1) — panic and short loss of consciousness due to not receiving enough oxygen
seizure (Nervous system disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECoG (electrocorticography) sensing (N=6)
Numbness in ear cup (Nervous system disorders) | 1 (1)
Decreased medical fitness (General disorders) | 1 (1)
High blood pressure, high heart rate and fever (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension, anemia and thrombocytopenia (General disorders) | 1 (1)
High inflammatory values (Infections and infestations) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1) — Temporary partial hearing loss in both ears after radiation therapy for excess saliva
pain in the neck (Musculoskeletal and connective tissue disorders) | 1 (2)
Occasional jaw lock (Musculoskeletal and connective tissue disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) — Blister on heel
Bladder infection (Renal and urinary disorders) | 1 (2)
Lower well being (General disorders) | 1 (1) — Lower emotional/psychological well being

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT02224469/Prot_SAP_000.pdf